CLINICAL TRIAL: NCT00081796
Title: A Randomized, Open-Label, Phase III Study of RPR109881 IV Every 3 Weeks Versus Capecitabine (Xeloda) Tablets Twice Daily for 2 Weeks in 3-Week Cycles in Patients With Metastatic Breast Cancer Progressing After Taxanes and Anthracycline Therapy
Brief Title: Breast Cancer Trial of RPR109881 Versus Capecitabine in Male or Female Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6089; XRP9881B-3001; NCT00107406 (obsolete NCT alias)
Record Dates: First submitted 2004-04-20; First posted 2004-04-22 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Breast Cancer; Metastases
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — larotaxel; RPR 109881A; Capecitabine

INTERVENTIONS:
Drug: larotaxel (RPR109881, XRP9881)
Drug: capecitabine

SUMMARY:
The purpose of this clinical trial is to determine if RPR109881 is a better treatment than capecitabine (Xeloda) for advanced breast cancer in patients that no longer benefit from docetaxel and/or paclitaxel.

DETAILED DESCRIPTION:
All patients in this trial will receive either the investigational drug or capecitabine, a chemotherapy drug that is already approved to treat your disease. These drugs prevent tumor cells from dividing, so they may stop growing or die. The investigational drug in this clinical trial is a chemotherapy drug given through the vein once every three weeks. Patients who receive capecitabine will receive this drug by mouth for 14 days, every 21 days.

ELIGIBILITY:
Eligibility Criteria

In order to be eligible for this trial you must:

* Have a diagnosis of breast cancer that is now metastatic (meaning the cancer has spread beyond its original location) or a recurrence of the cancer in its original location that cannot be removed by surgery.
* Have received previous treatment with anthracyclines (e.g., adriamycin, Doxorubicin) and taxanes (e.g., paclitaxel, docetaxel, Taxol®, Taxotere®) for your breast cancer and your doctor has determined that these treatment are no longer of benefit to you.
* Be at least 18 years of age.
* Not be taking other treatments for your cancer at the time you enter this trial.
* Not be pregnant.

Additionally, there are other criteria for study entry that a doctor participating in this study will need to review in detail with you and clinical assessments may need to be performed (e.g., lab tests, CT scans).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2004-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression.

SECONDARY OUTCOMES:
Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (180):
- United States (82):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Burbank, California
  - Concord, California
  - Fountain Valley, California
  - Fresno, California
  - Fullerton, California
  - Gilroy, California
  - Long Beach, California
  - Los Angeles, California
  - Monterey Park, California
  - Northridge, California
  - Oxnard, California
  - Pomona, California
  - Porterville, California
  - Redondo Beach, California
  - San Diego, California
  - San Francisco, California
  - Santa Barbara, California
  - Soquel, California
  - Vista, California
  - New London, Connecticut
  - Newark, Delaware
  - Fort Lauderdale, Florida
  - Gainsville, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Lawrenceville, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Centralia, Illinois
  - Chicago, Illinois
  - Peoria, Illinois
  - Skokie, Illinois
  - Fort Wayne, Indiana
  - New Albany, Indiana
  - Danville, Kentucky
  - Hazard, Kentucky
  - Lexington, Kentucky
  - Lafayette, Louisiana
  - Shreveport, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Saint Joseph, Michigan
  - Southfield, Michigan
  - St Louis, Missouri
  - Billings, Montana
  - Hackensack, New Jersey
  - Nyack, New York
  - Utica, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Worthington, Ohio
  - Dunmore, Pennsylvania
  - Hershey, Pennsylvania
  - Kingston, Pennsylvania
  - Kttaning, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Richardson, Texas
  - Abingdon, Virginia
  - Arlington, Virginia
  - Kirkland, Washington
  - Spokane, Washington
  - Huntington, West Virginia
- Argentina (3):
  - Buenos Aires
  - Capital Federal
  - Santa Fe
- Australia (4):
  - Melbourne
  - Perth
  - St Leonards
  - Sydney
- Austria (2):
  - Bludesch
  - Vienna
- Brazil (2):
  - Sorocaba, São Paulo
  - São Paulo
- Canada (7):
  - St. John's, Newfoundland and Labrador
  - Lévis, Quebec
  - Québec, Quebec
  - Montreal
  - Ontario
  - Ottawa
  - Québec
- Chile (2):
  - Las Condes, Santiago
  - Santiago
- Colombia (3):
  - Bogotá
  - Cali Valle
  - Medellín
- Czechia (3):
  - Hradec Králové
  - Nora Ves Pod Plesi
  - Ostrava
- Finland (2):
  - Kemi
  - Oulu
- France (8):
  - Besançon
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Saint-Cloud
  - Saint-Herblain
- Germany (9):
  - Aschaffenburg
  - Berlin
  - Frankfurt
  - Halle
  - Heidelberg
  - Kiel
  - Munchen Bayern
  - Munich
  - Oldenberg
- Hungary (2):
  - Budapest
  - Szeged
- Israel (5):
  - Ashkelon
  - Beersheba
  - Haifa
  - Tel Aviv
  - Tel Litwinsky
- Italy (10):
  - Bologna
  - Cuneo
  - Largo Agostino Gemelli
  - Livorno
  - Modena
  - Napoli
  - Novara
  - Palermo
  - Pavia
  - Sassari
- Mexico (2):
  - Mexico DF Distrio Federal
  - Tuluea Estand de Mexico
- New Zealand (2):
  - Auckland
  - Christchurch
- Poland (2):
  - Kracow
  - Warsaw
- Portugal (4):
  - Porto, Porto District
  - Beja
  - Coimbra
  - Lisbon
- Romania (3):
  - Bucharest, Bucharest
  - Cluj-Napoca
  - Craiova
- Maribor, Slovenia
- South Africa (5):
  - Capetown
  - Durban
  - Johannesburg
  - Parktown
  - Pretoria
- South Korea (2):
  - Gyeonggi-do
  - Seoul
- Spain (5):
  - Alicante
  - Jaén
  - Madrid
  - Navarra
  - Valencia
- Taiwan (2):
  - Taipai
  - Taoyuang
- United Kingdom (8):
  - Birmingham, Birmingham
  - Cardiff, Carduff
  - Bristol
  - Ipswich
  - London
  - Manchester
  - Nottingham
  - Surrey